CLINICAL TRIAL: NCT03883022
Title: Vancomycin Powder Combined With Autogenous Bone Graft as a Prevention for Post-operative Infection for Spine Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-10-008A
Record Dates: First submitted 2019-03-10; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Spinal Fusion; Spinal Stenosis; Spondylolisthesis
Keywords: Deep surgical site infection; Vancomycin-impregnated bone graft; Spine surgery; Degenerative lumbar disorder
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vancomycin (V Group) (Experimental)
  Interventions: Drug: with U-VANCO (vancomycin hydrochloride)
- Without Vancomycin (NV Group) (Active Comparator)
  Interventions: Drug: without U-VANCO (vancomycin hydrochloride)

INTERVENTIONS:
Drug: with U-VANCO (vancomycin hydrochloride) — 1 gm or 2 gm mixed with autogenous cancellous bone graft
  Arms: Vancomycin (V Group)
Drug: without U-VANCO (vancomycin hydrochloride) — no vancomycin added
  Arms: Without Vancomycin (NV Group)

SUMMARY:
Deep surgical site infection (DSSI) is one of the most challenging complications for spinal surgeons and can lead to a poor clinical outcome. This ambispective study was designed to examine the effect of vancomycin powder mixed with autogenous bone graft and bone substitute on preventing deep surgical site infection (DSSI) in degenerative lumbar fusion surgeries as well as any interference with bony fusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have instrumented spine fusion surgery due to failed conservative treatment (bed rest, medication, rehabilitation programs) for 3 to 6 months
* Patients who are willing to sign the surgical permit after the surgeon explains all surgical procedures along with the surgical risks
* Patients who fully understand the surgical procedures as well as the surgical risks and are willing to sign the surgical permit and the inform consent
* Patients who agree one more blood withdrawal after operation

Exclusion Criteria:

* Patients who agree to accept the spine surgery but do not agree to sign the inform consent
* Patients who have allergic reaction to vancomycin

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-09-03 (Actual); Primary Completion 2027-09-12 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Bony fusion status | Post-operative 1 month
  The bony fusion status (Lenke criteria)
Bony fusion status | Post-operative 3 months
  The bony fusion status (Lenke criteria)
Bony fusion status | Post-operative 6 months
  The bony fusion status (Lenke criteria)
Bony fusion status | Post-operative 1 year
  The bony fusion status (Lenke criteria)
Functional outcomes | Post-operative 1 month
  Functional outcomes, visual analogue scale (VAS)
Functional outcomes | Post-operative 3 months
  Functional outcomes, visual analogue scale (VAS)
Functional outcomes | Post-operative 6 months
  Functional outcomes, visual analogue scale (VAS)
Functional outcomes | Post-operative 1 year
  Functional outcomes,visual analogue scale (VAS)
Functional outcomes | Post-operative 1 months
  Functional outcomes,oswestry disability index (ODI)
Functional outcomes | Post-operative 3 months
  Functional outcomes, oswestry disability index (ODI)
Functional outcomes | Post-operative 6 months
  Functional outcomes, oswestry disability index (ODI)
Functional outcomes | Post-operative 1 year
  Functional outcomes, oswestry disability index (ODI)

SECONDARY OUTCOMES:
Vancomycin concentration | Post-operative days 1
  Vancomycin concentration was checked for both the serum and drainage.
Vancomycin concentration | Post-operative days 3
  Vancomycin concentration was checked for both the serum and drainage.

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Tien Wang, MD, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wang ST, Lin HH, Yao YC, Huang N, Hsiung W, Chang MC, Liu CL, Chou PH. Vancomycin powder mixed with autogenous bone graft and bone substitute may decrease the deep surgical site infections in elective lumbar instrumented fusion surgery for degenerative disorders: a prospective randomized study. Spine J. 2025 Sep;25(9):1866-1876. doi: 10.1016/j.spinee.2025.05.001. Epub 2025 May 5. PMID 40334989